CLINICAL TRIAL: NCT01817543
Title: A Multi-Center, Prospective, Cohort Trial Comparing the Effectiveness of AutoloGel Therapy to Usual and Customary Care in Venous Leg Ulcers
Brief Title: A Cohort Trial Comparing AutoloGel Therapy to Usual and Customary Care in Venous Leg Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol study design was re-done in collaboration with CMS
Sponsor: Cytomedix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM003
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Venous Leg Ulcer
Keywords: venous leg ulcers; non healing wounds
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AutoloGel (Experimental): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive Autologel treatment
  Interventions: Device: AutoloGel

INTERVENTIONS:
Device: AutoloGel — Autologel is a platelet-rich plasma gel used in the treatment of non-healing wounds
  Other Names: AutoloGel System

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, cohort-controlled trial in which venous leg ulcers (VLU)n will be treated using AutoloGel and case-matched against a concurrent cohort of patients receiving undefined Usual and Customary Care (UCC)

DETAILED DESCRIPTION:
Recurrence of ulcers in the leg is common; two-thirds of patients are likely to experience recurring ulcers after the first ulcer. While treatment of the underlying venous disease, depending on the mode of treatment, can lower the recurrence rate in many patients, it does not affect recurrence. AutoloGel is a platelet-rich plasma (PRP) gel used in the treatment of non-healing chronic wounds. The aim of this trial is to demonstrate the effectiveness, measured as complete wound healing, in a prospective, open-label trial in which venous leg ulcers will be treated using AutoloGel and standard of care and case-matched against a concurrent cohort of patients receiving undefined Usual and Customary Care

ELIGIBILITY:
Inclusion Criteria:

1. Medicare/Medicaid eligible
2. ≥18 years of age
3. Proven venous disease
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located between and including the knee and the ankle
5. For subjects with potentially multiple eligible VLUs, the largest ulcer will be selected. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 2 cm2 and 200 cm2
7. Demonstrated adequate compression regimen
8. Duration ≥ 1 month at first visit
9. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to AutoloGel components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Presence of another wound that is concurrently treated and might interfere with treatment of index wound by AutoloGel
3. Ulcer not of VLU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
4. Any malignancy other than non-melanoma skin cancer
5. Subjects who are cognitively impaired and do not have a healthcare proxy
6. Serum albumin of less than 2.5 g/dL
7. Plasma Platelet count of less than 100 x 109/L
8. Hemoglobin of less than 10.5 g/dL
9. Subject has inadequate venous access for repeated blood draw required for AutoloGel Administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to wound closure | 12 weeks
  Primary endpoint is time to wound healing after 12 weeks com pared with case matched controls receiving standard of care. Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart (FDA Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment, 2006).

SECONDARY OUTCOMES:
Proportion of wounds healed | 12 weeks
  Comparison of proportion of wounds healed over 12 weeks
Frequency of ulcer recurrence | 1 year
  Frequency of ulcer recurrence over a 1 year period post treatment; recurrence is defined as any new ulcer appearing on the leg after the index ulcer has healed.
Change in Quality of Life with Chronic Wounds (W-QOL) Score | 12 weeks
  Change in mean Quality of Life with Chronic Wounds (W-QOL) score between baseline and at 12 weeks
Number of patients with adverse events as a measure of tolerability | 12 weeks
  Frequency and severity of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arcadia, California
  - HyperBarxs at Northside Forsyth, Cumming, Georgia